CLINICAL TRIAL: NCT01260181
Title: Phase II, Open-Label Study of Erlotinib (Tarceva®) Treatment in Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer Who Present Activating Mutations in the Tyrosine Kinase Domain of the Epidermal Growth Factor Receptor
Brief Title: A Study of Erlotinib in Participants With Locally Advanced or Metastatic Non-Small Cell Lung Cancer With Epidermal Growth Factor Receptor Mutations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML25434; 2010-022509-17
Record Dates: First submitted 2010-12-13; First posted 2010-12-15 (Estimated); Results first posted 2018-10-26 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer
MeSH Terms: interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes

ARMS (1):
- Erlotinib (Experimental): Participants will receive erlotinib 150 millgrams (mg) orally daily until disease progression.
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Erlotinib — Erlotinib 150 mg tablet will be given orally daily.

SUMMARY:
This single arm, open-label study will evaluate the efficacy and safety of erlotinib (Tarceva) in participants with locally advanced or metastatic non-small cell lung cancer (NSCLC) with epidermal growth factor receptor (EGFR) mutations.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic NSCLC with EGFR mutations
* Measurable disease according to RECIST criteria
* Adequate hematological, renal and liver function

Exclusion Criteria:

* Previous chemotherapy or therapy against EGFR for metastatic disease
* Symptomatic cerebral metastases
* Pre-existing disease of the lung parenchyma such as lung fibrosis, lymphangitic carcinomatosis
* History of another malignancy except for carcinoma in-situ of the cervix, adequately treated basal cell skin carcinoma, or radically treated prostate carcinoma with good prognosis
* Concomitant use of coumarins

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-03-31 (Actual); Primary Completion 2017-09-29 (Actual); Study Completion 2017-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (9):
- Portugal (9):
  - Hospital Infante D. Pedro; Servico de Oncologia Medica, Aveiro
  - Hospital Geral; Servico de Pneumologia, Coimbra
  - IPO de Lisboa; Servico de Pneumologia, Lisbon
  - Hospital Santo Antonio dos Capuchos;Servico de Oncologia Medica, Lisbon
  - Hospital de Santa Maria; Servico de Pneumologia, Lisbon
  - Hospital Pulido Valente; Servico de Pneumologia, Lisbon
  - IPO do Porto; Servico de Oncologia Medica, Porto
  - Hospital de Sao Joao; Servico de Pneumologia, Porto
  - CHVNG/E_Unidade 1; Servico de Pneumologia, Vila Nova de Gaia

RESULTS

PARTICIPANT FLOW:
Groups:
- Erlotinib: Participants received erlotinib 150 millgrams (mg) orally daily until disease progression.
Period: Overall Study
Arm/Group | Erlotinib
Started | 30
Completed | 29
Not Completed | 1
Not completed — Decision of Investigator | 1

BASELINE CHARACTERISTICS:
Population: The intention to treat (ITT) population was defined as all subjects who are enrolled to the treatment phase of the study, regardless if they completed treatment.
Arm/Group | Erlotinib
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.33 (9.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 30

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Objective Response (Complete Response [CR]/Partial Response [PR]) Based on Computer Tomography (CT) or Magnetic Resonance Imaging (MRI) According to Response Evaluation Criteria in Solid Tumors (RECIST) Version (v) 1.1
Description: Objective response (OR) was based on criteria related to changes in size of target lesions according to modified RECIST. Target lesions were selected on the basis of their size (lesions with the longest diameter) as well as the feasibility of reproducible repeated measurements. OR was the sum of complete response (CR) and partial response (PR) four at least 4 weeks during treatment. CR: disappearance of all target lesions. PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: Baseline up to 5 years (assessed at Baseline, every 8 weeks until disease progression or death or end of treatment period [up to 5 years])
Population: The ITT population was defined as all subjects who are enrolled to the treatment phase of the study, regardless if they completed treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 30
percentage of participants | 63.3 [46.1 to 80.6]

2. Secondary Outcome: Progression Free Survival (PFS) Based on CT or MRI According to RECIST v 1.1
Description: Kaplan Meier estimate of the median PFS was defined as the time at which half of the participants have progressed (progressive disease [PD]) based on RECIST tumor response criteria or died from any cause, whichever occurred first. PD: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Patients who had not died or progressed at the time of the final analysis were censored at the date of last contact.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Erlotinib
Number analyzed (Participants) | 30
weeks | 40 [31 to 63]

3. Secondary Outcome: Overall Survival
Description: Overall Survival (OS) was defined as the time between the date of randomization and the date of death due to any cause.
Time Frame: Baseline up to 5 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Erlotinib
Number analyzed (Participants) | 30
weeks | 83 [56 to 125]

4. Secondary Outcome: Percentage of Participants With Adverse Events
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Baseline up to 5 years
Population: The safety population was identical to the ITT population, which included all participants enrolled in the study.
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 30
percentage of participants | 29

5. Secondary Outcome: Percentage of Participants With Epidermal Growth Factor Receptor (EGFR) Mutation in Study Population
Description: Mutations in the EGFR included exon 19 deletion mutations and the single-point substitution mutation L858R in exon 21.
Time Frame: Screening (21 days prior to Day 1)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 30
percentage of participants
  Exon 19 mutation | 40
  Exon 21 mutation | 60

6. Secondary Outcome: Median Time Taken From the First Response Until Disease Progression Based on RECIST v 1.1 as Determined by the Investigator
Description: The response duration was defined as the time of initial response (complete response (CR) /partial response (PR) whichever is first recorded) until documented disease progression. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial response was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Disease progression was defined as At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Erlotinib
Number analyzed (Participants) | 30
weeks | 41.5 [32 to 63]

ADVERSE EVENTS:
Time Frame: 5 years
Description: The safety population was identical to the ITT population, which included all participants enrolled in the study.
Arm/Group | Erlotinib
All-Cause Mortality (participants affected / at risk) | 4/30
Serious Adverse Events (participants affected / at risk) | 8/30
Other Adverse Events (participants affected / at risk) | 29/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=30)
Death (General disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Pneumonia (Infections and infestations) | 1
Intestinal Perforation (Gastrointestinal disorders) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Pelvic Infection (Infections and infestations) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Depression (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=30)
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 19
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 8
Alopecia (Skin and subcutaneous tissue disorders) | 5
Acne (Skin and subcutaneous tissue disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 15
Constipation (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 5
Stomatitis (Gastrointestinal disorders) | 5
Dyspepsia (Gastrointestinal disorders) | 3
Abdominal Pain (Gastrointestinal disorders) | 2
Odynophagia (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Paronychia (Infections and infestations) | 7
Upper Respiratory Tract Infection (Infections and infestations) | 7
Eye Infection (Infections and infestations) | 2
Conjunctivitis (Infections and infestations) | 6
Fatigue (General disorders) | 7
Oedema Peripheral (General disorders) | 5
Influenza Like Illness (General disorders) | 4
Asthenia (General disorders) | 3
Pain (General disorders) | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 5
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Bone Pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 2
Neck Pain (Musculoskeletal and connective tissue disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dry Eye (Eye disorders) | 5
Blepharitis (Eye disorders) | 2
Cataract (Eye disorders) | 2
Anxiety (Psychiatric disorders) | 4
Depression (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 3
Decreased Appetite (Metabolism and nutrition disorders) | 8
Hyperglycaemia (Metabolism and nutrition disorders) | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 2
Headache (Nervous system disorders) | 4
Dizziness (Nervous system disorders) | 3
Blood Bilirubin Increased (Investigations) | 2
Neutrophil Count Increased (Investigations) | 2
Weight Decreased (Investigations) | 2
Pollakiuria (Renal and urinary disorders) | 3
Leukocytosis (Blood and lymphatic system disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Statistical Analysis Plan (2014-03-28): https://cdn.clinicaltrials.gov/large-docs/81/NCT01260181/SAP_000.pdf
  • Study Protocol (2014-02-12): https://cdn.clinicaltrials.gov/large-docs/81/NCT01260181/Prot_001.pdf